CLINICAL TRIAL: NCT01181765
Title: The Efficacy of Open Label Infliximab for the Induction and Maintenance of Mucosal Healing in Small Bowel Crohn's Disease Assessed Through Wireless Camera Endoscopy (the ICE Study)
Brief Title: The Efficacy of Open Label Infliximab for the Induction and Maintenance of Mucosal Healing in Small Bowel Crohn's Disease Assessed Through Wireless Camera Endoscopy
Acronym: ICE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100747; P05088 (Other: Janssen Inc.)
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; infliximab; capsule endoscopy
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infliximab infusions (5 mg/kg) at weeks 0, 2, 6, 14 and 22 (Experimental)
  Interventions: Biological: Infliximab 5 mg/kg body weight infused over 2 hours

INTERVENTIONS:
Biological: Infliximab 5 mg/kg body weight infused over 2 hours — Subjects will receive IV Infusion of infliximab 5 mg/kg body weight at Week 0, Week 2, Week 6, Week 14 and Week 22 as per the approved Canadian product monograph of infliximab.

SUMMARY:
This is a pilot study to estimate the efficacy of infliximab in inducing and maintaining healing of lesions in the mucosa of subjects with Crohn's disease involving their small bowel.

DETAILED DESCRIPTION:
Landmark trials in Crohn's disease demonstrated the efficacy of infliximab in inducing and maintaining clinical remission. Furthermore, the endoscopic sub-studies within these trials demonstrated the ability of infliximab to rapidly induce and maintain mucosal healing as evidenced by the complete absence of mucosal breaks in the colon and terminal ileum. Unfortunately, conventional colonoscopy does not allow intestinal exploration beyond a very restricted portion of the small bowel (at most 10-15 cm of the terminal ileum). A study that systematically examines the changes in the small bowel mucosa during Crohn's disease symptomatic improvement is clearly needed.

This study consists of 20 subjects and 30 weeks of follow up. All subjects will undergo wireless camera endoscopy at three (3) visits, namely: at Screening, at Week 10 and at Week 26. Infliximab is administered at (5) visits, namely: at Baseline (week 0), Week 2, Week 6, Week 14 and Week 22. In some subjects, an ileal-colonoscopy may be performed at Week 26.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Established diagnosis of Crohn's disease and evidence of small bowel involvement
* CDAI score between 220 and 450 inclusively
* Lewis score of at least 790 at Screening
* Colonoscopy within the last 6 months
* Successful excretion of the intact patency capsule Exclusion Criteria
* Contraindications to anti-TNF therapy (TB, cardiac impairment, etc.)
* Prior bowel resection
* Prior anti-TNF exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Endoscopic Improvement | Week 26
  Mean change in Lewis score between Baseline and Week 26

SECONDARY OUTCOMES:
Clinical improvement | Week 26
  Mean change in Crohn's Disease Activity Index (CDAI) between Baseline and Week 26.
Early endoscopic improvement | Week 10
  Mean change in Lewis score between Baseline and Week 10
Clinical Improvement | Week 10
  Mean change in CDAI between Baseline and Week 10

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Inc. Clinical Trial, Study Director — Janssen Inc.
Locations (2):
- Canada (2):
  - Ottawa, Ontario
  - Toronto, Ontario

REFERENCES:
- See also: The Efficacy of Open-Label Infliximab for the Induction and Maintenance of Mucosal Healing in Small Bowel Crohn's Disease Assessed Through Wireless Camera Endoscopy (the ICE study). — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3412&filename=CR100747_CSR.PDF